CLINICAL TRIAL: NCT05082558
Title: Clinical Characteristics and Prognostic Factors of Atrial Fibrillation at a Tertiary Center of Pakistan - From a South-Asian Lens - a Retrospective Study.
Status: Completed | Type: Observational
Sponsor: Aga Khan University Hospital, Pakistan (Other)
Responsible Party: Principal Investigator, Pirbhat Shams, Dr. Pirbhat Shams, Resident, Adult Cardiology, Department of Medicine, The Aga Khan University, Aga Khan University Hospital, Pakistan
Other Study IDs: 2019-1008-2905
Record Dates: First submitted 2021-09-07; First posted 2021-10-19 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention, as this was retrospective study. — No intervention performed. Participants were entolled retrospectively and medical records were accessed for data.

SUMMARY:
To evaluate the clinical characteristics and management purseued for atrial fibrillation in a tertiary care center of Pakistan. We aimed at looking baseline characteristics and associated co-morbid conditions and primary diagnosis associated with atrial fibrillation.

DETAILED DESCRIPTION:
It is a retrospective observational study done at Aga Khan University Hospital, Karachi, Pakistan, which is a tertiary care teaching hospital with a cardiology and cardiac surgery center. Aga Khan Hospital is one of the main referral health centers in Pakistan.

This study was approved by Aga Khan University ethical review committee (ERC No. # 2019-1008-2905).We reviewed hospital record files of 651 patients including both males and females, admitted in Aga Khan University Hospital from 1st July 2018 to 31st December 2018, who were found to have atrial fibrillation as a primary or associated diagnosis. Diagnosis of atrial fibrillation was confirmed on a 12 lead ECG. Fifteen patients were excluded who did not have electrocardiographic evidence of atrial fibrillation.

For all patient, demographic information including age and gender, reason of admission and duration of arrhythmia were noted from the written medical records. Comorbidities were tabulated including: diabetes mellitus, hypertension, coronary artery disease, heart failure, cardiomyopathy, valvular heart disease, chronic obstructive pulmonary disease, and hyperthyroidism. Echocardiographic data were reviewed for left atrial (LA) dimension, LA volume index and left ventricular (LV) systolic function.

Patients were labeled as Diabetic if they had HbA1c of >6.5gm/dl or they were already on treatment for diabetes mellitus. Hypertension was defined as average of two readings of systolic blood pressure of ≥140mmHg or diastolic blood pressure of ≥90mmHg or patients already taking antihypertensive medications. Coronary artery disease was defined as ≥50% stenosis in at least one of the epicardial coronary arteries. Cardiomyopathy was defined as left ventricular ejection fraction of ≤50% Chronic obstructive pulmonary disease was defined as forced expiratory volume in 1st second to forced vital capacity ratio of <70% of the predicted value. Patients were labeled hyperthyroid if they have low serum TSH and high serum concentration of free T4 or T3 as per laboratory reference range.

All patients were followed from the time of inclusion to the time of discharge or till inpatient death. Hemodynamic parameters including heart rate and blood pressure were recorded at the time of inclusion for patients with known atrial fibrillation and at the time of onset of arrhythmia for those with new onset atrial fibrillation. Patients' treatment record were reviewed for medications. Complications related to atrial fibrillation or its treatment were recorded.

ELIGIBILITY:
Inclusion Criteria:

* inpatients
* Age >/= 18 years
* Having atrial fibrillation on 12 lead surface EKG.
* Both males and females.

Exclusion Criteria:

* Age <18 years.
* Non-availability of 12 lead EKG.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We reviewed hospital record files of 651 patients including both males and females, admitted in Aga Khan University Hospital from 1st July 2018 to 31st December 2018, who were found to have atrial fibrillation as a primary or associated diagnosis. Diagnosis of atrial fibrillation was confirmed on a 12 lead ECG.
Sampling Method: Non-Probability Sample
Enrollment: 651 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Clinical charcateristics and management features of atrial fibrillation | July 2018 to December 2018
  To evaluate baseline characteristics of patients admitted with atrial fibrillation.

SECONDARY OUTCOMES:
Clinical charcateristics of atrial fibrillation patients | July 2018 to December 2018
  To identify and compare clinical characteristics of patients with atrial fibrillation.

CONTACTS AND LOCATIONS:
Locations (1):
- The Aga Khan University, Karachi, Pakistan